CLINICAL TRIAL: NCT00918983
Title: Phase III Multicenter Prospective Randomized Parallel-Group Placebo-Controlled Double Blind Clinical Evaluation of NX-1207 for the Treatment of BPH NX02-0017
Brief Title: Clinical Evaluation of NX-1207 for the Treatment of Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nymox Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NX02-0017
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign prostatic hyperplasia; BPH; Enlarged prostate
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — fexapotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NX-1207 (Experimental)
  Interventions: Drug: NX-1207
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NX-1207 — Single intraprostatic injection of 2.5 mg NX-1207
  Arms: NX-1207
Drug: Placebo — Single intraprostatic injection of placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of a 2.5 mg dose of NX-1207 for the treatment of BPH (benign prostatic hyperplasia) as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed informed consent prior to enrolment in the study
2. IPSS ≥ 15
3. Prostate Volume ≥ 30 mL ≤ 70 mL
4. Qmax < 15 mL/sec based on a minimum void of 125 mL
5. Agree not to use any other approved or experimental BPH or OAB medication anytime during the study

Exclusion Criteria:

1. History of illness or condition that may interfere with study or endanger subject
2. Use of prescribed medications that may interfere with study or endanger subject
3. Presence of a median lobe of the prostate
4. Previous surgery or MIST for treatment of BPH
5. Post-void residual urine volume > 200 mL
6. PSA ≥ 10 ng/mL; prostate cancer must be ruled out (negative biopsy) for PSA ≥ 4 ng/mL
7. Participation in a study of any investigational drug or device within the previous 90 days
8. Prostate cancer

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2009-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) | 365 days

SECONDARY OUTCOMES:
International Prostate Symptom Score (IPSS) | 90 days
International Prostate Symptom Score (IPSS) | 180 days
International Prostate Symptom Score (IPSS) | 270 days
Peak urine flow rate (Qmax) | 365 days
Peak urine flow rate (Qmax) | 90 days
Peak urine flow rate (Qmax) | 180 days

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - For information concerning this clinical site, please contact Nymox at 800-936-9669, Birmingham, Alabama
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Huntsville, Alabama
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Tucson, Arizona
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Little Rock, Arkansas
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Anaheim, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Atherton, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., La Mesa, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Long Beach, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Los Alamitos, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Denver, Colorado
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., New Britain, Connecticut
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Naples, Florida
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Ocala, Florida
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Orlando, Florida
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Tallahassee, Florida
  - For information concerning this clinical site, please contact Nymox at 800-936-9669, Atlanta, Georgia
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Roswell, Georgia
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Forest Hill, Indiana
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Jeffersonville, Indiana
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Shreveport, Louisiana
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Missoula, Montana
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Lawrenceville, New Jersey
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Mount Laurel, New Jersey
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Voorhees Township, New Jersey
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Brooklyn, New York
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Garden City, New York
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Poughkeepsie, New York
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Concord, North Carolina
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Raleigh, North Carolina
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Cincinnati, Ohio
  - For information concerning this clinical site, please contact Nymox at 800-936-9669, Columbus, Ohio
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Bethany, Oklahoma
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Salem, Oregon
  - For information concerning this clinical site, please contact Nymox at 800-936-9669, Bala-Cynwyd, Pennsylvania
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Lancaster, Pennsylvania
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Myrtle Beach, South Carolina
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Knoxville, Tennessee
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Arlington, Texas
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Carrollton, Texas
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Dallas, Texas
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Salt Lake City, Utah